CLINICAL TRIAL: NCT03922451
Title: Pharmacokinetics of Antibiotics During Extracorporeal Membrane Oxygenation (ECMO) Support
Status: Terminated | Type: Observational
Why Stopped: COVID-19 - study and recruitment not feasible
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Katie Moynihan, Cardiac Intensivist, Boston Children's Hospital
Other Study IDs: IRB-P00030970
Record Dates: First submitted 2019-04-15; First posted 2019-04-22 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Drug Effect
MeSH Terms: interventions — Piperacillin, Tazobactam Drug Combination; Cefazolin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pediatric patients supported on ECMO
  Interventions: Drug: piperacillin-tazobactam; Drug: Cefazolin

INTERVENTIONS:
Drug: piperacillin-tazobactam — Administered for infection treatment or prophylaxis per hospital protocol
Drug: Cefazolin — Administered for infection treatment or prophylaxis per hospital protocol

SUMMARY:
This study will measure plasma concentrations of piperacillin-tazobactam and cefazolin in pediatric patients supported with extracorporeal membrane oxygenation (ECMO) aiming to better understand the pharmacokinetics of these medications in this in vivo setting.

ELIGIBILITY:
Inclusion Criteria:

* supported on ECMO
* receive piperacillin-tazobactam or cefazolin as part of routine care or infection management

Exclusion Criteria:

* >= 18 years
* No Consent provided

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All pediatric patients who are supported on ECMO at Boston Children's Hospital Cardiac Intensive Care Unit (CICU) and receive piperacillin-tazobactam or cefazolin as part of routine care or infection management.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2019-08-27 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Plasma concentration: piperacillin-tazobactam | Peri drug dose administration until cessation of antibiotic therapy or cessation of ECMO support up to a maximum of 4 weeks.
  Drug levels will be checked at baseline followed by additional measurements after the dose based on the dosing intervals but anticipated to be 30, 60, 120, 360, 480 minutes after the dose. Dosing regime will be q8-12 hourly pending end organ function (at the discretion of the treating team). The study will be continued for the duration of the Antibiotic therapy whilst on ECMO support and for one set of samples following decannulation.
Plasma concentration: cefazolin | Peri drug dose administration until cessation of antibiotic therapy or cessation of ECMO support up to a maximum of 4 weeks.
  Drug levels will be checked at baseline followed by additional measurements after the dose based on the dosing intervals but anticipated to be 30, 60, 120, 360, 480 minutes after the dose. Dosing regime will be q8-12 hourly pending end organ function (at the discretion of the treating team). The study will be continued for the duration of the Antibiotic therapy whilst on ECMO support and for one set of samples following decannulation.

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States